CLINICAL TRIAL: NCT07260110
Title: TEPLIzumab: QUality of Life Evaluation During Stage Transition
Brief Title: A Longitudinal, Observational Study Comparing Real-World Experiences of Teplizumab-Treated and Untreated Participants With Stage 2 Type 1 Diabetes in the United States
Acronym: TEPLI-QUEST
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS18679; U1111-1319-0170 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-10-29; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — teplizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with a history of teplizumab infusion: Participants with a history of stage 2 type 1 diabetes who have been infused with teplizumab at the time of enrollment
  Interventions: Drug: Teplizumab
- Participants with no history of teplizumab infusion: Participants with stage 2 type 1 diabetes who have not been infused with teplizumab at the time of enrollment

INTERVENTIONS:
Drug: Teplizumab — This study will not administer any treatment, only observe the treatment as prescribed in real-world clinical practice.
  Other Names: TZIELD
  Groups: Participants with a history of teplizumab infusion

SUMMARY:
This study is an observational, longitudinal, non-interventional real-world study in the United States. The study is meant to describe the experience of participants with a history of stage 2 type 1 diabetes who have been infused with teplizumab and the experience of participants with stage 2 type 1 diabetes who have not been infused with teplizumab, and to compare descriptively the experiences of the two groups.

Primary Objective:

- To characterize health related quality of life, diabetes-related anxiety, diabetes-related burden, and ease of diabetes management, and how participants feel, form and function in those who infused and those who did not infuse with teplizumab

Secondary Objectives:

* To show the clinical transitions experienced by those who infused and those who did not infuse with teplizumab
* To describe the prevalence and timing of diabetes misclassification and the temporal patterns between misclassification, antibody testing, and the correct diagnosis of type 1 diabetes in those who infused and those who did not infuse with teplizumab
* To estimate the impact of diagnostic misclassification on the timing of progression to stage 3 type 1 diabetes in those who infused and those who did not infuse with teplizumab
* To characterize glucose monitoring strategies in those who infused and those who did not infuse with teplizumab where possible
* To characterize insulin use in those who infused and those who did not infuse with teplizumab where possible
* To characterize longitudinal health care resource utilization in those who infused and those who did not infuse with teplizumab

DETAILED DESCRIPTION:
Each participant is expected to participate in the study from the time of their enrollment through the last data delivery, which is estimated to occur five years after the first participant is enrolled.

ELIGIBILITY:
Inclusion Criteria:

* History of stage 2 type 1 diabetes with the presence of one or more diabetes-related autoantibodies and dysglycemia confirmed in the medical record
* At the time of enrollment either not yet diagnosed with stage 3 type 1 diabetes, or the progression occurred in the last 18 months prior to enrollment
* Aged 8 or older at the time of enrollment
* Aged 8 or older at the time of teplizumab infusion (if infused)
* Receipt of medical care in the United States
* Able to and does give written informed consent

Exclusion Criteria:

- Failure to complete the baseline survey

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a history of Stage 2 T1D (documented in medical records) and infused with teplizumab or not infused with teplizumab
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2030-12-03 (Estimated); Study Completion 2030-12-03 (Estimated)

PRIMARY OUTCOMES:
Change in participant and caregiver-reported outcomes from survey responses: ease of diabetes management questions | From baseline, repeated every 6 months up to end of study, approximately 5 years
Change in participant and caregiver-reported outcomes from survey responses: Psychological well-being World Health Organization-5 (WHO-5) | From baseline, repeated every 6 months up to end of study, approximately 5 years
Change in participant and caregiver-reported outcomes from survey responses: State-Trait Anxiety Inventory (STAI) | From baseline, repeated every 6 months up to end of study, approximately 5 years
Change in participant and caregiver-reported outcomes from survey responses: Type 1 Diabetes Distress Assessment System-Core Scale (T1-DDAS CORE) | From baseline, repeated every 6 months, up to end of study, approximately 5 years
Change in participant and caregiver-reported outcomes from survey responses: Diabetes constraints scale | From baseline, repeated every 6 months up to end of study, approximately 5 years
Sociodemographic screening characteristics | At enrollment
Sociodemographic medical history characteristics | At enrollment
Sociodemographic diabetes management characteristics | At enrollment

SECONDARY OUTCOMES:
Changes in characteristics of participants: monitoring practices (e.g. continuous glucose monitor, self-monitoring blood glucose, blood drawn by clinician) across type 1 diabetes stages | From enrollment up to study end, approximately 5 years
Changes in characteristics of participants: medical history across type 1 diabetes stages | From enrollment up to study end, approximately 5 years
Time from index date to the diagnosis of stage 3 type 1 diabetes | From baseline up to end of study, approximately 5 years
Changes in glucose parameters: HbA1c | From baseline up to end of study, approximately 5 years
Changes in glucose parameters: blood glucose | From baseline up to end of study, approximately 5 years
Changes in glucose parameters: post prandial glucose | From baseline up to end of study, approximately 5 years
Changes in glucose parameters: c-peptide | From baseline up to end of study, approximately 5 years
Changes in glucose parameters: time in range in participants with glucose monitor data | From baseline up to end of study, approximately 5 years
Changes in glucose parameters: time above range in participants with glucose monitor data | From baseline up to end of study, approximately 5 years
Changes in glucose parameters: time below range in participants with glucose monitor data | From baseline up to end of study, approximately 5 years
Changes in glucose parameters: glucose variability percent in participants with glucose monitor data | From baseline up to end of study, approximately 5 years
Changes in glucose parameters: percent coefficient of variation in participants with glucose monitor data | From baseline up to end of study, approximately 5 years
Changes in glucose paremeters: glucose management indicator in participants with glucose monitor data | From baseline up to end of study, approximately 5 years
Number of complications (including micro- and macrovascular occurrences and hypoglycemia occurrences) | From baseline up to end of study, approximately 5 years
The frequency of glycemic vs. autoantibody testing related to stage 2 type 1 diabetes diagnosis | At enrollment
The sequence (first or second) of glycemic testing vs. autoantibody testing related to stage 2 type 1 diabetes diagnosis | At enrollment
  Sequence describes if glycemic testing or autoantibody testing took place first in stage 2 type 1 diabetes diagnosis
The frequency of misclassification with type 2 diabetes | At enrollment
The time between misclassification with type 2 diabetes and autoantibody testing | At enrollment
The time between misclassification with type 2 diabetes and the correct diagnosis of stage 2 type 1 diabetes | At enrollment
Time from index date to the diagnosis of stage 3 type 1 diabetes for those misclassified with type 2 diabetes where diagnosis is confirmed by HbA1c and/or glycemic measures | From baseline up to end of study, approximately 5 years
Proportion (%) of participants using home glycemic monitoring assessments (Continuous Glucose Monitor, self-monitoring blood glucose, urine glucose monitoring) vs in-clinic assessments (HbA1c, fasting blood glucose, c-peptide) | From baseline up to end of study, approximately 5 years
Proportion (%) of participants using insulin characterized by insulin dosing, type, regimen, and mode of administration | From baseline up to end of study, approximately 5 years
Annualized rate of hospitalizations due to type 1 diabetes complications | From baseline up to end of study, approximately 5 years
Annualized rate of emergency room visits due to type 1 diabetes complications | From baseline up to end of study, approximately 5 years
Annualized rate of specialist (including endocrinologist) visits | From baseline up to end of study, approximately 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Site, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: OBS18679 Tepli-QUEST website for potential participants — https://picnichealth.com/care/programs/tepli-quest